CLINICAL TRIAL: NCT03970694
Title: Neoadjuvant Chemoradiotherapy Versus Neoadjuvant Chemotherapy For Unresectable Locally Advanced Colon Cancer: An Open, Multi-centered, Randomize Controlled Phase 3 Trial.
Brief Title: Neoadjuvant Chemoradiotherapy Versus Neoadjuvant Chemotherapy For Unresectable Locally Advanced Colon Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Significant differences in conversion rate as well as R0 resection rate between the two groups.
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Fujian Medical University Union Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Nanfang Hospital, Southern Medical University (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Yuan-hong Gao, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-FXY-194
Record Dates: First submitted 2019-05-26; First posted 2019-05-31 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Colon Cancer
Keywords: Neoadjuvant chemoradiotherapy; Colon Cancer; Initial Diagnosed Unresectable Locally Advanced Stage; Phase 3 Clinical Trial
MeSH Terms: conditions — Colonic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Research group: Neoadjuvant chemoradiotherapy group Control group: Neoadjuvant chemotherapy group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant chemoradiotherapy group (Experimental): Neoadjuvant chemoradiotherapy（XELOX * 4 + radiotherapy）→ Surgery (if possible) → post-surgery chemotherapy.
  Interventions: Radiation: Radiotherapy; Drug: oxaliplatin+capecitabine
- Neoadjuvant chemotherapy group (Other): Arm Type: control. Neoadjuvant chemotherapy（XELOX * 4）→ Surgery (if possible) → post-surgery chemotherapy.
  Interventions: Drug: oxaliplatin+capecitabine

INTERVENTIONS:
Radiation: Radiotherapy — Since 2006, neoadjuvant chemoradiotherapy has been a recommendation as standard treatment for locally advanced rectal cancer, and has been widely applied to clinical use. As for locally advanced colon cancer, it still lacks evidence to support whether neoadjuvant chemoradiotherapy is a beneficial option.We recently reported clinical data about therapeutic effect of 60 unresectable locally advanced colon cancer cases and it was exciting. According to our results, through neoadjuvant chemoradiotherapy, R0 resection rate is 86%, local recurrence rate is 10.2%, 3-year OS and 5-year OS are 76.7% and 66.6%, respectively."Colorectal cancer diagnoses and treatment guidelines" written by Chinses Society of Clinical Oncology (ver. 2017, 2018), suggested that neoadjuvant chemoradiotherapy was an optional treatment strategy or secondary recommended treatment strategy.
  Arms: Neoadjuvant chemoradiotherapy group
Drug: oxaliplatin+capecitabine — Colorectal cancer is one of the most common malignant tumors, the morbidity and mortality rate are both in rising trend. 10-23% newly diagnosed colon cancer is at locally advanced stage and surgical unresectable. For this subgroup, treatment guidelines recommend neoadjuvant chemotherapy with or without targeted therapy.

SUMMARY:
A. Background and purpose:

Neoadjuvant chemoradiotherapy versus neoadjuvant chemotherapy for unresectable locally advanced colon cancer: an open, multi-centered, randomize controlled phase 3 trial.

Colorectal cancer is one of the most common malignant tumors, the morbidity and mortality rate are both in rising trend. 10-23% newly diagnosed colon cancer is at locally advanced stage and surgically unresectable. For this subgroup, treatment guidelines recommend neoadjuvant chemotherapy with or without targeted therapy. However, less than 50% patients could convert into R0 resectable, therapeutic effect is unsatisfactory, 5-year overall survival rate is only 12.5%-45.7%.[JCO,2010] Since 2006, neoadjuvant chemoradiotherapy has been a recommendation as standard treatment for locally advanced rectal cancer, and has been widely applied to clinical use. As for locally advanced colon cancer, it still lacks evidence to support whether neoadjuvant chemoradiotherapy is a beneficial option. There are only several articles about locally advanced colon cancer undertaking neoadjuvant chemoradiotherapy before surgery through Pubmed research, including 3 case reports, 1 abstract and 5 clinical researches with a small sample size, 3 of which are from the investigator's study group.

The investigators recently reported clinical data about therapeutic effect of 60 unresectable locally advanced colon cancer cases and the results were exciting. According to the results, through neoadjuvant chemoradiotherapy, R0 resection rate is 86%, local recurrence rate is 10.2%, 3-year OS and 5-year OS are 76.7% and 66.6%, respectively. [Onco Targets Ther, 2018] "Colorectal cancer diagnoses and treatment guidelines" written by Chinses Society of Clinical Oncology (ver. 2017, 2018), suggested that neoadjuvant chemoradiotherapy was an optional treatment strategy or secondary recommended treatment strategy. In a word, the investigators' result was referred as revisory basis of the guideline [CJC,2016], with a relatively low level of evidence in evidence-based medicine.

This phase 3 clinical trial mainly aims to acquire a higher level of evidence in evidence-based medicine on the subject about neoadjuvant chemoradiotherapy as a treatment strategy to unresectable locally advanced colon cancer, and the ultimate goal is to rewrite the International treatment guidelines of locally advanced colorectal cancer.

B. Research Content:

1. . Research Object: Patients who newly diagnosed unresectable locally advanced colon cancer. Including: 1. tumor infiltrates through the intestinal wall and adheres to tissues and organs around the colon(T4b), imaging assesses that R0 resection is unachievable. 2. Pericolonic lymph node involvement is closely adjacent to the large abdominal vessels, imaging assesses that lymphadenectomy is difficult. 3. Surgical exploration indicates that R0 resection is not achievable. 4. In initial diagnosis, surgeon evaluates the need for extensive multi-organ combined resection and expected to damage the organs, which would seriously affect the postoperative quality of life.
2. . Main research indicator: 5-year overall survival rate
3. . Secondary research indicators: 1. R0 resection rate 2. 3-year tumor-free survival rate
4. . Research groups assignment: 1. Research group: Neoadjuvant chemoradiotherapy group; 2. Control group: Neoadjuvant chemotherapy group.
5. . Sample calculation: Calculation is based on the main research indicator: 5-year survival rate. Based on α=0.05(bilateral), β=0.20(unilateral), 5-year OS improves from 45% in control group to 65% in research group, 4-year period, 5-year follow-up. Research group and control group should at least enroll 74 and 75 qualified cases, respectively, a total of 149 cases, with an expected delisting rate of 20%, the total sample size is 186, 93 cases for each group.
6. . Research protocols:

1. Research group: Neoadjuvant chemoradiotherapy（XELOX * 4 + radiotherapy）→ Surgery (if possible) → post-surgery chemotherapy.

2. Control group: Neoadjuvant chemotherapy（XELOX * 4）→ Surgery (if possible) → post-surgery chemotherapy.

Chemotherapy strategy: XELOX: oxaliplatin 130mg/m2, iv drip, d1, every 3 weeks; capecitabine 1,000mg/m2, bid, d1-d14, every 3 weeks. Concurrent chemotherapy: mXELOX: which oxaliplatin is 100mg/m2.

Radiotherapy strategy: IMRT, 6-8MV X-ray; GTV 45-50Gy/25F, 1.8-2.0Gy/F; CTV 42.5-45Gy/25F, 1.7-1.8Gy/F; Actual delivery dose should be adjusted according to max tolerance dose of organs at risk, but the delivery dose of GTV and CTV must within the required range.

Surgery: Reexamination is performed 5 weeks after radiotherapy for research group and 2 weeks after the fourth period of chemotherapy, surgery is performed in 6-12 weeks after neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histology confirms colonic adenocarcinoma.
* The distance from the lower edge of the tumor to the anal edge is greater than or equal to 15cm (from sigmoid colon to ileocecal region)
* Preoperative staging (Satisfying any one out of four conditions below)

  1. Tumor infiltrates through the intestinal wall and adheres to tissues and organs around the colon(T4b), imaging assesses that R0 resection is unachievable.
  2. Pericolonic lymph node involvement is closely adjacent to the large abdominal vessels, imaging assesses that lymphadenectomy is difficult.
  3. Surgical exploration indicates that R0 resection is not achievable.
  4. In initial diagnosis, surgeon evaluates the need for extensive multi-organ combined resection and expected to damage the organs, which would seriously affect the postoperative quality of life.
* No obvious signs of intestinal obstruction, or obstruction has been relieved after proximal enterostomy.
* Preoperative CT/MRI/PET-CT has ruled out distant metastasis.
* Blood and biochemical indexes achieve standard (Satisfying all three conditions below):

  1. Routine blood test: WBC>4000/mm3; PLT>100000/mm3; Hb>6g/dl.
  2. Liver function: SGOT, SGPT and Bilirubin are less than or equal to 1.5 times normal upper limit.
  3. Renal function: Creatinine is less than or equal to 1.5 times normal upper limit.

Exclusion Criteria:

* History: Has colon surgery history; Received chemotherapy or biotherapy in the past 5 years; Received radiotherapy in treatment field.
* Infectious disease: HIV infection history; Active phase chronic hepatitis B or hepatitis C (high copies of virus DNA); Other serious active clinical infection.
* Diagnosed as stage I colon cancer.
* Extraperitoneal distant metastasis is positive in pre-operative stage.
* Dyscrasia or organ decompensation.
* Received radiation therapy in abdominal or pelvic regions.
* Multiple primary cancer.
* Epileptic seizures requiring medical treatment.
* Other malignant tumor history in the past 5 years (except endocervical cancer in situ or skin basal cell carcinoma which had been cured)
* Chronic inflammatory colorectal disease, unrelieved ileus.
* Drug abuse, has medical, psychological or social condition that might affect research results.
* Allergic to research-related drugs.
* Any unstable situation that might endanger patient's safety or compliance.
* Pregnant, lactating woman patient or fertile but lacks adequate contraceptives.
* Refuses to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-05-11 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
5-year overall survival rate | 5 years after treatment
  The percentage of patients survive 5 years after treatment.

SECONDARY OUTCOMES:
R0 resection rate | an average of 6 to 12 weeks after surgery
  The percentage of patients whose post-operative pathology indicate negative margin is observed under microscope
3-year progression-free survival rate | 3 years after treatment
  The percentage of patients have no tumor progression after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-hong Gao, M.D, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Curley SA, Carlson GW, Shumate CR, Wishnow KI, Ames FC. Extended resection for locally advanced colorectal carcinoma. Am J Surg. 1992 Jun;163(6):553-9. doi: 10.1016/0002-9610(92)90554-5. PMID 1595834
- [Background] Eldar S, Kemeny MM, Terz JJ. Extended resections for carcinoma of the colon and rectum. Surg Gynecol Obstet. 1985 Oct;161(4):319-22. PMID 4049200
- [Background] Lehnert T, Methner M, Pollok A, Schaible A, Hinz U, Herfarth C. Multivisceral resection for locally advanced primary colon and rectal cancer: an analysis of prognostic factors in 201 patients. Ann Surg. 2002 Feb;235(2):217-25. doi: 10.1097/00000658-200202000-00009. PMID 11807361
- [Background] Croner RS, Merkel S, Papadopoulos T, Schellerer V, Hohenberger W, Goehl J. Multivisceral resection for colon carcinoma. Dis Colon Rectum. 2009 Aug;52(8):1381-6. doi: 10.1007/DCR.0b013e3181ab580b. PMID 19617748
- [Background] Govindarajan A, Coburn NG, Kiss A, Rabeneck L, Smith AJ, Law CH. Population-based assessment of the surgical management of locally advanced colorectal cancer. J Natl Cancer Inst. 2006 Oct 18;98(20):1474-81. doi: 10.1093/jnci/djj396. PMID 17047196
- [Background] Reibetanz J, Germer CT. [Neoadjuvant chemotherapy for locally advanced colon cancer : Initial results of the FOxTROT study.]. Chirurg. 2013 Oct 13. doi: 10.1007/s00104-013-2631-8. Online ahead of print. No abstract available. German. PMID 24122133
- [Background] Karoui M, Koubaa W, Delbaldo C, Charachon A, Laurent A, Piedbois P, Cherqui D, Tran Van Nhieu J. Chemotherapy has also an effect on primary tumor in colon carcinoma. Ann Surg Oncol. 2008 Dec;15(12):3440-6. doi: 10.1245/s10434-008-0167-9. Epub 2008 Oct 11. PMID 18850249
- [Background] Foxtrot Collaborative Group. Feasibility of preoperative chemotherapy for locally advanced, operable colon cancer: the pilot phase of a randomised controlled trial. Lancet Oncol. 2012 Nov;13(11):1152-60. doi: 10.1016/S1470-2045(12)70348-0. Epub 2012 Sep 25. PMID 23017669
- [Background] Arredondo J, Pastor C, Baixauli J, Rodriguez J, Gonzalez I, Vigil C, Chopitea A, Hernandez-Lizoain JL. Preliminary outcome of a treatment strategy based on perioperative chemotherapy and surgery in patients with locally advanced colon cancer. Colorectal Dis. 2013 May;15(5):552-7. doi: 10.1111/codi.12119. PMID 23398577
- [Background] Arredondo J, Gonzalez I, Baixauli J, Martinez P, Rodriguez J, Pastor C, Ribelles MJ, Sola JJ, Hernandez-Lizoain JL. Tumor response assessment in locally advanced colon cancer after neoadjuvant chemotherapy. J Gastrointest Oncol. 2014 Apr;5(2):104-11. doi: 10.3978/j.issn.2078-6891.2014.006. PMID 24772338
- [Background] Masi G, Loupakis F, Salvatore L, Fornaro L, Cremolini C, Cupini S, Ciarlo A, Del Monte F, Cortesi E, Amoroso D, Granetto C, Fontanini G, Sensi E, Lupi C, Andreuccetti M, Falcone A. Bevacizumab with FOLFOXIRI (irinotecan, oxaliplatin, fluorouracil, and folinate) as first-line treatment for metastatic colorectal cancer: a phase 2 trial. Lancet Oncol. 2010 Sep;11(9):845-52. doi: 10.1016/S1470-2045(10)70175-3. Epub 2010 Aug 9. PMID 20702138
- [Background] Loupakis F, Cremolini C, Masi G, Lonardi S, Zagonel V, Salvatore L, Cortesi E, Tomasello G, Ronzoni M, Spadi R, Zaniboni A, Tonini G, Buonadonna A, Amoroso D, Chiara S, Carlomagno C, Boni C, Allegrini G, Boni L, Falcone A. Initial therapy with FOLFOXIRI and bevacizumab for metastatic colorectal cancer. N Engl J Med. 2014 Oct 23;371(17):1609-18. doi: 10.1056/NEJMoa1403108. PMID 25337750
- [Background] Yamada Y, Takahari D, Matsumoto H, Baba H, Nakamura M, Yoshida K, Yoshida M, Iwamoto S, Shimada K, Komatsu Y, Sasaki Y, Satoh T, Takahashi K, Mishima H, Muro K, Watanabe M, Sakata Y, Morita S, Shimada Y, Sugihara K. Leucovorin, fluorouracil, and oxaliplatin plus bevacizumab versus S-1 and oxaliplatin plus bevacizumab in patients with metastatic colorectal cancer (SOFT): an open-label, non-inferiority, randomised phase 3 trial. Lancet Oncol. 2013 Dec;14(13):1278-86. doi: 10.1016/S1470-2045(13)70490-X. Epub 2013 Nov 11. PMID 24225157
- [Background] de Gramont A, Van Cutsem E, Schmoll HJ, Tabernero J, Clarke S, Moore MJ, Cunningham D, Cartwright TH, Hecht JR, Rivera F, Im SA, Bodoky G, Salazar R, Maindrault-Goebel F, Shacham-Shmueli E, Bajetta E, Makrutzki M, Shang A, Andre T, Hoff PM. Bevacizumab plus oxaliplatin-based chemotherapy as adjuvant treatment for colon cancer (AVANT): a phase 3 randomised controlled trial. Lancet Oncol. 2012 Dec;13(12):1225-33. doi: 10.1016/S1470-2045(12)70509-0. Epub 2012 Nov 16. PMID 23168362
- [Background] Taieb J, Tabernero J, Mini E, Subtil F, Folprecht G, Van Laethem JL, Thaler J, Bridgewater J, Petersen LN, Blons H, Collette L, Van Cutsem E, Rougier P, Salazar R, Bedenne L, Emile JF, Laurent-Puig P, Lepage C; PETACC-8 Study Investigators. Oxaliplatin, fluorouracil, and leucovorin with or without cetuximab in patients with resected stage III colon cancer (PETACC-8): an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Jul;15(8):862-73. doi: 10.1016/S1470-2045(14)70227-X. Epub 2014 Jun 11. PMID 24928083
- [Background] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Background] Gerard JP, Conroy T, Bonnetain F, Bouche O, Chapet O, Closon-Dejardin MT, Untereiner M, Leduc B, Francois E, Maurel J, Seitz JF, Buecher B, Mackiewicz R, Ducreux M, Bedenne L. Preoperative radiotherapy with or without concurrent fluorouracil and leucovorin in T3-4 rectal cancers: results of FFCD 9203. J Clin Oncol. 2006 Oct 1;24(28):4620-5. doi: 10.1200/JCO.2006.06.7629. PMID 17008704
- [Background] Bosset JF, Collette L, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Ollier JC; EORTC Radiotherapy Group Trial 22921. Chemotherapy with preoperative radiotherapy in rectal cancer. N Engl J Med. 2006 Sep 14;355(11):1114-23. doi: 10.1056/NEJMoa060829. PMID 16971718
- [Background] Roh MS, Colangelo LH, O'Connell MJ, Yothers G, Deutsch M, Allegra CJ, Kahlenberg MS, Baez-Diaz L, Ursiny CS, Petrelli NJ, Wolmark N. Preoperative multimodality therapy improves disease-free survival in patients with carcinoma of the rectum: NSABP R-03. J Clin Oncol. 2009 Nov 1;27(31):5124-30. doi: 10.1200/JCO.2009.22.0467. Epub 2009 Sep 21. PMID 19770376
- [Background] Hallet J, Zih FS, Lemke M, Milot L, Smith AJ, Wong CS. Neo-adjuvant chemoradiotherapy and multivisceral resection to optimize R0 resection of locally recurrent adherent colon cancer. Eur J Surg Oncol. 2014 Jun;40(6):706-12. doi: 10.1016/j.ejso.2014.01.009. Epub 2014 Feb 2. PMID 24534363
- [Background] Kuga Y, Tanaka T, Arita M, Okanobu H, Miwata T, Yoshimi S, Murakami E, Numata Y, Moriya T, Ohya T, Nishida T. [A case of effective chemotherapy using S-1 and CPT-11 following chemoradiotherapy with UFT and Leucovorin for unresectable advanced sigmoid colon cancer]. Gan To Kagaku Ryoho. 2010 Mar;37(3):531-4. Japanese. PMID 20332698
- [Background] Yoh T, Yamamichi K, Oishi M, Iwaki R, Motohiro T. [A case of effective neoadjuvant chemoradiotherapy with capecitabine for locally advanced sigmoid colon cancer]. Gan To Kagaku Ryoho. 2011 Jun;38(6):1021-4. Japanese. PMID 21677500
- [Background] Yoshitomi M, Hashida H, Nomura A, Ueda S, Terajima H, Osaki N. [A case of locally advanced sigmoid colon cancer treated with neoadjuvant chemoradiotherapy]. Gan To Kagaku Ryoho. 2014 Sep;41(9):1175-8. Japanese. PMID 25248907
- [Background] Burton S, Brown G, Daniels I, Norman A, Swift I, Abulafi M, Wotherspoon A, Tait D. MRI identified prognostic features of tumors in distal sigmoid, rectosigmoid, and upper rectum: treatment with radiotherapy and chemotherapy. Int J Radiat Oncol Biol Phys. 2006 Jun 1;65(2):445-51. doi: 10.1016/j.ijrobp.2005.12.027. PMID 16690432
- [Background] O'Neill B, Brown G, Wotherspoon A, Burton S, Norman A, Tait D. Successful downstaging of high rectal and recto-sigmoid cancer by neo-adjuvant chemo-radiotherapy. Clin Med Oncol. 2008;2:135-44. doi: 10.4137/cmo.s348. Epub 2008 Mar 1. PMID 21892276
- [Background] Cukier M, Smith AJ, Milot L, Chu W, Chung H, Fenech D, Herschorn S, Ko Y, Rowsell C, Soliman H, Ung YC, Wong CS. Neoadjuvant chemoradiotherapy and multivisceral resection for primary locally advanced adherent colon cancer: a single institution experience. Eur J Surg Oncol. 2012 Aug;38(8):677-82. doi: 10.1016/j.ejso.2012.05.001. Epub 2012 May 24. PMID 22632848
- [Background] Qiu B, Ding PR, Cai L, Xiao WW, Zeng ZF, Chen G, Lu ZH, Li LR, Wu XJ, Mirimanoff RO, Pan ZZ, Xu RH, Gao YH. Outcomes of preoperative chemoradiotherapy followed by surgery in patients with unresectable locally advanced sigmoid colon cancer. Chin J Cancer. 2016 Jul 7;35(1):65. doi: 10.1186/s40880-016-0126-y. PMID 27389519
- [Background] Chang H, Yu X, Xiao WW, Wang QX, Zhou WH, Zeng ZF, Ding PR, Li LR, Gao YH. Neoadjuvant chemoradiotherapy followed by surgery in patients with unresectable locally advanced colon cancer: a prospective observational study. Onco Targets Ther. 2018 Jan 17;11:409-418. doi: 10.2147/OTT.S150367. eCollection 2018. PMID 29398921
- [Derived] Zhang ZT, Xiao WW, Li LR, Wu XJ, Wang QX, Chang H, Tian X, Jiang W, Lin JZ, Zhang RX, Fan WH, Pan ZZ, Zhang R, Gao YH. Neoadjuvant chemoradiotherapy versus neoadjuvant chemotherapy for initially unresectable locally advanced colon cancer: short-term outcomes of an open-label, single-centre, randomised, controlled, phase 3 trial. EClinicalMedicine. 2024 Sep 21;76:102836. doi: 10.1016/j.eclinm.2024.102836. eCollection 2024 Oct. PMID 39364270